CLINICAL TRIAL: NCT06462027
Title: A Single-center, Randomized, Placebo Controlled Pilot Study of Packed Red Blood Cell Transfusion During Prolonged Adult In-hospital Cardiac Arrest
Brief Title: Packed Red Blood Cell Transfusion During Cardiac Arrest
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 18-01273
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Packed Red Blood Cells (1 unit) (Experimental): 500 mL of packed red blood cells
  Interventions: Drug: Packed Red Blood Cells (1 unit)
- Packed Red Blood Cells (2 units) (Experimental): 1000 mL of packed red blood cells
  Interventions: Drug: Packed Red Blood Cells (2 units)
- Saline solution (Placebo Comparator): Treatment of 500 mL of normal saline.
  Interventions: Other: Saline

INTERVENTIONS:
Drug: Packed Red Blood Cells (1 unit) — 500 mL of packed red blood cells administered intravenously 10-20 minutes after CA onset, provided Return of Spontaneous Circulation (ROSC) has not been achieved.
  Arms: Packed Red Blood Cells (1 unit)
Drug: Packed Red Blood Cells (2 units) — 1000 mL of packed red blood cells administered intravenously 10-20 minutes after CA onset, provided Return of Spontaneous Circulation (ROSC) has not been achieved.
  Arms: Packed Red Blood Cells (2 units)
Other: Saline — Control subjects will receive 500mL of normal saline intravenously.
  Arms: Saline solution

SUMMARY:
The purpose of this pilot interventional study is to collect preliminary data on administering packed red blood cell (PRBC) during cardiac arrest (CA). The primary objective is to assess the feasibility of PRBC transfusion during cardiac CA to help optimize the methods required to augment cerebral and other vital organ oxygen delivery during cardiopulmonary resuscitation (CPR). The secondary objectives are to assess the effect of PRBC transfusion during prolonged cardiac arrests on cerebral oxygenation, end tidal carbon dioxide (ETCO2), return of spontaneous circulation (ROSC), survival to discharge, biomarkers of neural injury and inflammation, and neurological outcomes at hospital discharge, 30 days post-CA, and 90 days post-CA.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age ≥18 and <85 years
* Experience prolonged, non-trauma-related in-hospital cardiac arrest, defined by cessation of heartbeat and respiration requiring CPR for at least 10 minutes

Exclusion Criteria:

* Age <18 years old
* Age > 85 years old
* Patients with DNR/DNI orders (Do Not Resuscitate/Do Not Intubate)
* Patients admitted to the hospital with a cardiac arrest arising from trauma
* Patients who achieve return of spontaneous circulation within 10 minutes of CPR
* Inability to start study product administration within 20 minutes of cardiac arrest onset
* Prisoners
* Women who are known to be pregnant
* Patients with a history of RBC antibodies or positive antibody screen prior to enrollment in the study, unless previously cross-matched units are available for transfusion.
* Patients with ultrasound evidence of right ventricular dilatation at time of CA
* Patients with known prior objection to receipt of blood products.
* Patients for whom administration of additional fluid volume is contraindicated (as determined by physician responsible for care)
* Physician objection based on concern that intervention would interfere with patient care plan

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Time (in mins) to administration of Packed Red Blood Cells (PRBC) | During Cardiopulmonary Resuscitation (CPR) (up to 20 minutes)
Frequency of antibody-mediated transfusion reactions | 6-72 hours after Return of Spontaneous Circulation (ROSC)
  Outcome measure will be evaluated for the occurrence of intravascular and extravascular hemolytic reactions by measuring fibrinogen, D-dimer, platelet count, peripheral blood smear, and serum haptoglobin.
Frequency of non-immune reactions | 6-72 hours after ROSC
  Non-immune reactions include Transfusion Associated Circulatory Overload (TACO) and Transfusion-Related Acute Lung Injury (TRALI) as determined by the Data Safety Monitoring Committee (DSMC).
Change in frequency of right ventricular (RV) dilatation | Baseline, up to 20 minutes post administration of PRBC
All-cause mortality | Up to 30 days after the last day of study participation
  Mortality due to all causes
Proportion of patients with unfavorable neurological outcomes | Up to 30 days post-Cardiac Arrest (CA)
  The Cerebral Performance Category (CPC) score is a five-point scale used to assess neurological outcome after cardiac arrest and other events. Scores range from 1 to 5, a score of 1 or 2 is considered a favorable outcome, and scores of 3, 4, or 5 are considered an unfavorable outcome (severe neurological disability, persistent vegetative state or death).

SECONDARY OUTCOMES:
Absolute change in peak regional oxygen saturation (rSO2) | 2 minutes prior to administration, 5 minutes post administration of PRBC
Absolute change in mean rSO2 | 2 minutes prior to administration, 5 minutes post administration of PRBC
Relative change in peak rSO2 | 2 minutes prior to administration, 5 minutes post administration of PRBC
Relative change in mean rSO2 | 2 minutes prior to administration, 5 minutes post administration of PRBC
Relative change in peak end tidal carbon dioxide (ETCO2) | 2 minutes prior to administration, 5 minutes post administration of PRBC
Relative change in mean ETCO2 | 2 minutes prior to administration, 5 minutes post administration of PRBC
Rate of ROSC | During CPR (up to 20 minutes)
Proportion of patients with release of pro-inflammatory cytokines | 6-72 hours after ROSC
Proportion of patients with release markers of brain injury | 6-72 hours after ROSC
Rate of survival | At time of hospital discharge (approximately 12 days)
Rate of survival | 30 days post-CA
Rate of survival | 90 days post-CA
CPC score | At time of hospital discharge (approximately 12 days)
  The Cerebral Performance Category (CPC) score is a five-point scale used to assess neurological outcome after cardiac arrest and other events. Scores range from 1 to 5, a score of 1 or 2 is considered a favorable outcome, and scores of 3, 4, or 5 are considered an unfavorable outcome (severe neurological disability, persistent vegetative state or death).
CPC score | 30 days post-CA
  The Cerebral Performance Category (CPC) score is a five-point scale used to assess neurological outcome after cardiac arrest and other events. Scores range from 1 to 5, a score of 1 or 2 is considered a favorable outcome, and scores of 3, 4, or 5 are considered an unfavorable outcome (severe neurological disability, persistent vegetative state or death).
CPC score | 90 days post-CA
  The Cerebral Performance Category (CPC) score is a five-point scale used to assess neurological outcome after cardiac arrest and other events. Scores range from 1 to 5, a score of 1 or 2 is considered a favorable outcome, and scores of 3, 4, or 5 are considered an unfavorable outcome (severe neurological disability, persistent vegetative state or death).

CONTACTS AND LOCATIONS:
Overall Officials: Sam Parnia, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Sam.Parnia@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data upon reasonable request. Requests should be directed to Sam.Parnia@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.